CLINICAL TRIAL: NCT03437395
Title: Accelerated Partial Breast Irradiation Study for Women With Stage 0 or 1 Breast Cancer
Brief Title: Accelerated Partial Breast Irradiation Study
Acronym: APBI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sentara Norfolk General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09.01
Record Dates: First submitted 2018-01-03; First posted 2018-02-19 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer Female
Keywords: Lumpectomy; Unifocal Disease; Stage 0 or 1 Disease

STUDY DESIGN:
Intervention Model Description: Patients will be offered either balloon brachytherapy or 3D conformal radiation therapy to treat the tumor bed alone. Data will be collected so that our results can be compared to the results of the randomized trial. Specifically, we will be comparing our local control rates and cosmetic results to those of favorable risk patients from the NSABP B-39 trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Partial Breast Irradiation (Other): All participants will be treated with partial breast irradiation by utilizing 3D conformal external beam irradiation or balloon brachytherapy. This is not a randomized study.
  Interventions: Device: Balloon Brachytherapy; Radiation: 3D Conformal External Beam Irradiation

INTERVENTIONS:
Device: Balloon Brachytherapy — The balloon brachytherapy catheter method uses one tube with a small balloon on the end placed where the tumor had been. The balloon is filled with salt water so it fits this space. The end of the tube will extend from the side of the breast and will be connected to a special machine for treatments. The RT dose is delivered by a radioactive seed that travels through the tube into the center of the balloon. The seed will be removed at the end of each treatment. The tube and the balloon filled with salt water will stay in the breast until the 10 RT treatments are done. The radiation oncologist will decide if this type of treatment is most appropriate for the patient. The treatment will be given 2 times a day, about 6 hours apart, on 5 days. Each treatment lasts for 10-15 minutes.
Radiation: 3D Conformal External Beam Irradiation — 3D conformal external beam irradiation uses a beam of radiation to deliver the radiation therapy dose to the place in the breast where the cancer was removed. The Radiation Oncologist will decide which type of treatment is most appropriate for the patient. The treatment will be given 2 times a day, about 6 hours apart, on 5 days. Each treatment lasts for 10 to 15 minutes.

SUMMARY:
Breast cancer patients at Sentara RMH Hahn Cancer Center who are treated with accelerated partial breast irradiation will be monitored over a period of 10 years. From this group of patients, local and regional recurrence rates will be determined. Patients in the registry will also take part in assessments of cosmesis and quality of life.

DETAILED DESCRIPTION:
Studies have shown that giving radiation therapy to the breast after lumpectomy helps keep cancer from coming back in the breast. The purpose of this study is to see if partial breast irradiation (PBI) at SRMH Hahn Cancer Center is as good as partial breast irradiation performed in other centers in the United States in keeping cancer from coming back in the breast. Whole breast irradiation (WBI) is a standard treatment after a lumpectomy. WBI is radiation therapy given 5 days a week for 5 to 7 weeks to the whole breast. PBI is a new method of delivering radiation only to the area of the breast where the cancer was removed. PBI is given 2 times a day for 5 days. PBI may be given over a period of 5 to 10 days. This newer treatment is currently being compared with WBI in a randomized trial. Thus far, patients at low risk for cancer recurrence who have been treated with PBI have had excellent outcomes at 5 years post-treatment, but we will not know for sure if PBI is as good as WBI until the results of the randomized trial are available. However, PBI is commonly being offered outside of clinical trials in many community hospitals throughout the country. As radiation oncologists at Sentara RMH Hahn Cancer Center, we wanted to offer patients in our community the same opportunity to have this treatment, but also wanted to ensure close follow-up of all patients treated with this method, to be sure our results are similar to those of patients reported in our professional literature. There are two different methods of PBI that are being used at SRMH Hahn Cancer Center: Balloon brachytherapy and 3-D conformal external beam irradiation. This study will learn about the good and bad effects of radiation therapy. The study also will learn about the feelings women have about how their breast looks after surgery and radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* The patient must consent to be in the study and must have signed an approved consent form approved by Sentara RMH Medical Center's IRB.
* Patients must be >/= 50 years or postmenopausal.
* The patient must have stage 0 or 1 breast cancer.
* On histological examination, the tumor must be DCIS or invasive non- lobular carcinoma of the breast.
* Surgical treatment of the breast must have lumpectomy. The margins of the resected specimen must be histologically free of tumor (DCIS and in- vasive) by 2 mm or more. Reexcision of surgical margins is permitted.
* Gross disease must be unifocal with pathologic (invasive and/or DCIS) tumor size 2 cm or less. Mucinous or tubular histologies maximum size may be up to 3 cm.
* Patients with invasive breast cancer are required to have axillary staging which can include sentinel node biopsy alone (if sentinel node is negative), sentinel node biopsy followed by axillary dissection or sampling with a minimum total of 6 axillary nodes including the sentinel nodes (if sentinel node is positive), or axillary dissection alone (with a minimum of 6 axillary nodes.) (Axillary staging is not required for patients with DCIS).
* The patient must begin treatment within 9 weeks following the last surgery for breast cancer (lumpectomy, re-excision of margins, or axillary staging procedure).
* Patients must have an estrogen receptor (ER) and progesterone receptor (PR) analysis performed on the primary tumor prior to enrollment.
* The target lumpectomy cavity must be clearly delineated and the ratio of target lumpectomy cavity/whole breast reference volume must be </= 25% based on the postoperative CT scan.
* Patients are eligible if, based on the postoperative CT scan, PBI is judged to be technically deliverable by either 3D conformal radiation therapy or balloon brachytherapy.
* At the time of study entry, patients must have had an H&P within 4 months and a bilateral mammogram within 6 months.
* Patients with a history of non-breast malignancies are eligible if they have been disease-free for 5 or more years prior to study entry and are deemed by their physician to be low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, carcinoma in situ of the colon, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.

Exclusion Criteria: Men are not eligible for this study. Women with one or more of the following conditions are ineligible for this study.

* Stage II, Stage III, or Stage IV Breast Cancer
* Histologically positive axillary on non-axillary nodes.
* Palpable or radiographically suspicious ipsilateral or contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes, unless there is histologic confirmation that these nodes are negative for tumor.
* Suspicious microcalcifications, densities, or palpable abnormalities (in the ipsilateral or contralateral breast) unless biopsied and found to be benign.
* Non-epithelial breast malignancies such as sarcoma or lymphoma.
* Proven multicentric carcinoma (invasive or DCIS) in more than one quadrant or separated by 4 or more cm.
* Paget's disease of the nipple.
* Synchronous bilateral invasive or non-invasive breast cancer.
* History of invasive breast cancer or DCIS in the ipsilateral breast (Patients with a history of LCIS treated by surgery alone are eligible).
* Surgical margins that cannot be microscopically assessed or are less than 2 mm at pathologic evaluation. (if surgical margins are rendered free of disease by re-excision, the patient is eligible).
* Clear delineation of the extent of the target lumpectomy cavity not possible.
* Treatment plan that includes regional nodal irradiation.
* Any treatment with radiation therapy to the ipsilateral breast, chemo- therapy biotherapy, and/or hormonal therapy administered for the currently diagnosed breast cancer prior to study. The only exception is hormonal therapy, which may have been given for no more than a total of 28 days anytime after diagnosis and before study entry. For patients receiving chemotherapy, hormonal therapy must stop at or before study entry and resume following completion of chemotherapy. For patients not receiving chemotherapy, hormonal therapy may continue.
* Current therapy with any hormonal agents such as raloxifere (Evista), tamoxifen, or other selective receptor modulators (SERMs), either for osteoporosis or breast cancer prevention (patients are eligible only if these medications are discontinued prior to study entry).
* Breast implants. (Patients who have implants removed are eligible)
* Prior ipsilateral breast or thoracic RT for any condition.
* Collagen vascular disease, specifically dermatomyositis with CPK level above normal or with an active skin rash, systemic lupus erythematosis, or scleroderma.
* Pregnancy or lactation at the time of proposed study entry. Women of reproductive potential must agree to use an effective non-hormonal method of contraception during therapy.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who satisfy all of the eligibility conditions are the only patients who will be eligible for this study.
Enrollment: 139 (Actual)
Dates: Start 2009-03-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Local and Regional Recurrence after Partial Breast Irradiation as assessed by change in Physical Exam, Mammography, MRI, Scintimammography, Biopsy, and/or Surgical Pathology. | Prior to radiation, 4 weeks post RT, 6 months post RT, then yearly up to 10 1/2 years Post RT
  At the time of analysis, recurrence rates in the study group will be compared to recurrence rates in stage 1 breast cancer patients with similar risk factors from the national studies of APBI and whole breast radiation therapy, to determine if SRMH recurrence rates are significantly different.

SECONDARY OUTCOMES:
Number of Participants with Certain Characteristics or Risk Factors in SRMH Population that are Associated with a Higher Risk for Recurrence when Using Partial Breast Irradiation as Assessed by History and Physical, Mammography, Pathology. | prior to radiation, 4 weeks post RT, 6 months post RT, then yearly up to 10 1/0 years post RT
  At the time of analysis, it will also be determined whether these characteristics or risk factors in SRMH population are associated with a higher risk for recurrence when using this technique.

OTHER OUTCOMES:
Number of Participants will have Cosmetic Results Assessed by Utilizing the Breast Cancer Treatment Outcome Scale (BCTOS) using Patient Self Reports and a Cosmetic Evaluation Will Be Made by the Radiation Oncologist (or Surgeon). | Prior to radiation, 4 weeks post RT, 6 months post RT, then yearly up to 10 1/2 years post RT
  The patients will be monitored for cosmesis. Physician-generated versus patient-generated ratings will be compared to characterize the evaluation of cosmetic outcome from multiple perspectives. The Radiation Oncologist (or Surgeon) will utilize criteria established in previous RTOG trials.
Number of Participants will have Quality of Life Results Assessed by Utilizing the Breast Cancer Treatment Outcome Scale (BCTOS) using Patient Self Reports for Global Quality of Life. | Prior to radiation, 4 weeks post RT, 6 months post RT, then yearly up to 10 1/2 years
  The Breast Cancer Treatment Outcome Scale ( BCTOS) will be used as a primary measure to assess breast-related symptoms and treatment effects. Questionnaires will be used from the current RTOG trial of PBI vs. WBI to assess these measures using Patient Self Reports for Global Quality of Life. In evaluating the difference between the treated and untreated breast and area, the patient will select from none (assigned a value of 1, slight (assigned a value of 2), moderate (assigned a value of 3), and large (assigned a value of 4). Higher value indicates a larger difference between treated and untreated breast and area, which would be considered a worse outcome.
Number of Participants will have Fatigue Results Assessed by Utilizing the Breast Cancer Treatment Outcome Score (BCTOS) using Patient Self Reports. | Prior to radiation, 4 weeks post RT, 6 months post RT, then yearly up to 10 1/2 years.
  The Medical Outcomes Study Short Form-36 ( MOS SF-36 Vitality Scale), a widely used measure with high reliability and validity, will assess fatigue. The patient will select how much of the time during the past four weeks did she feel full of life, have a lot of energy, feel worn out, and feel tired. There are five values that include all the time (assigned a value of 1), most of the time (assigned a value of 2), some of the time (assigned a value of 3), a little of the time (assigned a value of 4), and none of the time (assigned a value of 5). Full of life and have a lot of energy,a low number would be the better outcome and feel worn out and feel tired, higher number would be the better outcome.
Number of Participants will have Treatment Related Symptoms Assessed by Utilizing the Breast Cancer Treatment Outcome Scale (BCTOS) using Patient Self Reports. | Prior to radiation, 4 weeks post RT, 6 months post RT, then yearly up to 10 1/2 years
  The Breast Cancer Treatment Outcome Score ( BCTOS) has been augumented with a brief set of additional items that focus specifically on radiotherapy-relevant symptoms (e.g., reports of skin problems, tenderness in the breast, hardness in the breast due to enhanced fibrosis, and pain). These questions relate to how much the patient has been bothered by these radiotherapy-relevant symptoms in the past four weeks. The patient will select from not bothered at all (assigned a score of 0), a little bit bothered (assigned a score of 1), somewhat bothered (assigned a score of 2), bothered quite a bit (assigned a score of 3), and bothered very much (assigned a score of 4.) The total value range is 0-92. Higher value indicates worse outcome.
Number of Participants will have Convenience of Care Assessed by Utilizing the Breast Cancer Treatment Outcome Scale (BCTOS) using Patient Self Reports | Prior to radiation, 4 weeks post RT, 6 months post RT, then yearly up to 10 1/2 years
  The Convenience of Care scale includes several items designed to assess how disruptive the treatment is on the patients' daily activities and life styles, as well as how satisfied the patients are with the duration of their treatment. By circling one number on a scale from 0 (not at all bothered) up to 10 (bothered quite a lot. Total value range is 0-80. The higher the value, the worse the outcome. The patient will evaluate her satisfaction about the treatment and results by selecting the phrase that best describes her satisfaction from totally satisfied (assigned a value of 1, somewhat satisfied (assigned a value of 2), neither satisfied or dissatisfied (assigned a value of 3), somewhat dissatisfied (assigned a value of 4), and totally dissatisfied (assigned a value of 5). The higher the value, the worse the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Heather A. Morgan, MD, Principal Investigator — Sentara RMH Medical Center
Locations (1):
- Sentara RMH Hahn Cancer Center, Harrisonburg, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher B, Anderson S, Bryant J, Margolese RG, Deutsch M, Fisher ER, Jeong JH, Wolmark N. Twenty-year follow-up of a randomized trial comparing total mastectomy, lumpectomy, and lumpectomy plus irradiation for the treatment of invasive breast cancer. N Engl J Med. 2002 Oct 17;347(16):1233-41. doi: 10.1056/NEJMoa022152. PMID 12393820
- [Background] Fisher ER, Dignam J, Tan-Chiu E, Costantino J, Fisher B, Paik S, Wolmark N. Pathologic findings from the National Surgical Adjuvant Breast Project (NSABP) eight-year update of Protocol B-17: intraductal carcinoma. Cancer. 1999 Aug 1;86(3):429-38. doi: 10.1002/(sici)1097-0142(19990801)86:33.0.co;2-y. PMID 10430251
- [Background] EORTC Breast Cancer Cooperative Group; EORTC Radiotherapy Group; Bijker N, Meijnen P, Peterse JL, Bogaerts J, Van Hoorebeeck I, Julien JP, Gennaro M, Rouanet P, Avril A, Fentiman IS, Bartelink H, Rutgers EJ. Breast-conserving treatment with or without radiotherapy in ductal carcinoma-in-situ: ten-year results of European Organisation for Research and Treatment of Cancer randomized phase III trial 10853--a study by the EORTC Breast Cancer Cooperative Group and EORTC Radiotherapy Group. J Clin Oncol. 2006 Jul 20;24(21):3381-7. doi: 10.1200/JCO.2006.06.1366. Epub 2006 Jun 26. PMID 16801628
- [Background] Polgar C, Fodor J, Major T, Nemeth G, Lovey K, Orosz Z, Sulyok Z, Takacsi-Nagy Z, Kasler M. Breast-conserving treatment with partial or whole breast irradiation for low-risk invasive breast carcinoma--5-year results of a randomized trial. Int J Radiat Oncol Biol Phys. 2007 Nov 1;69(3):694-702. doi: 10.1016/j.ijrobp.2007.04.022. Epub 2007 May 25. PMID 17531400
- [Background] Chao KK, Vicini FA, Wallace M, Mitchell C, Chen P, Ghilezan M, Gilbert S, Kunzman J, Benitez P, Martinez A. Analysis of treatment efficacy, cosmesis, and toxicity using the MammoSite breast brachytherapy catheter to deliver accelerated partial-breast irradiation: the william beaumont hospital experience. Int J Radiat Oncol Biol Phys. 2007 Sep 1;69(1):32-40. doi: 10.1016/j.ijrobp.2007.02.026. Epub 2007 Apr 30. PMID 17467920
- [Background] Vicini FA, Remouchamps V, Wallace M, Sharpe M, Fayad J, Tyburski L, Letts N, Kestin L, Edmundson G, Pettinga J, Goldstein NS, Wong J. Ongoing clinical experience utilizing 3D conformal external beam radiotherapy to deliver partial-breast irradiation in patients with early-stage breast cancer treated with breast-conserving therapy. Int J Radiat Oncol Biol Phys. 2003 Dec 1;57(5):1247-53. doi: 10.1016/s0360-3016(03)01573-6. PMID 14630258
- [Background] Haffty BG, Vicini FA, Beitsch P, Quiet C, Keleher A, Garcia D, Snider H, Gittleman M, Zannis V, Kuerer H, Whitacre E, Whitworth P, Fine R, Keisch M. Timing of Chemotherapy after MammoSite radiation therapy system breast brachytherapy: analysis of the American Society of Breast Surgeons MammoSite breast brachytherapy registry trial. Int J Radiat Oncol Biol Phys. 2008 Dec 1;72(5):1441-8. doi: 10.1016/j.ijrobp.2008.02.070. Epub 2008 Aug 7. PMID 18692330
- [Background] Martin Keish, M.D., Douglas Arthur, M.D., Rakesh Patel, M.D., Mark Rivard, PhD., Frank Vicini, M.D. February, 2007, American Brachytherapy Society Breast Brachytherapy Task Group. www.americanbrachytherapy.org/resources/abs_breast_brachytherapy_taskgroup.pdf
- [Background] NSABP B-39, RTOG 0413: A Randomized Phase III Study of conventional whole breast irradiation versus partial breast irradiation for women with stage 0, I, or II breast cancer. Clin Adv Hematol Oncol. 2006 Oct;4(10):719-21. No abstract available. PMID 17111558